CLINICAL TRIAL: NCT01831388
Title: Breath Training Exercise for the Reduction of Chronic Dyspnea: a Pilot Study
Brief Title: Breath Training Exercise for the Reduction of Chronic Dyspnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-261
Record Dates: First submitted 2013-04-08; First posted 2013-04-15 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Chronic Pulmonary Disorder
Keywords: Dyspnea; Breath Training Exercise; 12-261
MeSH Terms: conditions — Dyspnea

ARMS (1):
- The breath training program (Experimental): Approximately 30-minutes of group instruction session on breathing techniques delivered at a Main Campus outpatient clinic, followed by approximately 15 minutes twice daily home practice for six weeks with weekly telephone coaching. The intervention will conclude at about week 6. Patients will be encouraged to continue the practice, but there will be no further phone calls to remind patients or to confirm their continuing practice.
  Interventions: Other: breathing techniques; Behavioral: Self-Administered Baseline and Transition Dyspnea Indexes

INTERVENTIONS:
Other: breathing techniques — During all practice sessions, patients are seated in a chair, where they are guided through a set routine of various breathing techniques (detailed in Appendix A). No yoga poses are involved. There is no demand on the patient's physical condition and no risk of injury. The breath training program, with patients seated throughout, includes:
  - an initial teaching session (approximately 30-minute) at main campus by an MSKCC Integrative Medicine Service yoga-breathing instructor; - twice daily,breathing exercises (each approximately 15-minute) for 6 weeks practiced by patients at home with supplied recorded audio instructions; - and weekly follow-up phone calls by research staff (+/- 3 days from day 7 of each week) to identify and manage problems and to determine compliance.
Behavioral: Self-Administered Baseline and Transition Dyspnea Indexes — Patients are asked to complete baseline SAC-BDI/TDI questionnaires at the pulmonary clinic. Patients will return to the pulmonary clinic at about week 6 for SAC-BDI/TDI and tests, and to return the diary recording their home exercises. Resting and post-6MWT pulse oximetry, and Hospital Anxiety and Depression Scale (HADS) will be evaluated as well.

SUMMARY:
The purpose of this study is to test whether a breath training exercise program may be used to make patients with chronic lung conditions feel less short of breath, whether such a program is well received by patients and whether a future larger study is worthwhile.

The breath training exercise program uses some breathing techniques derived from Yoga practices. They were shown to help patients experiencing shortness of breath feel less short of breath in other settings. Whether the training is beneficial to patients with chronic lung conditions, especially those with a history of cancer affecting their lungs, is not clear. This study would help us answer that question.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of a chronic pulmonary disorder (a diagnosis of lung cancer is not required as the symptom of dyspnea, not cancer itself, is targeted)
* If diagnosed with lung cancer, must have completed definitive treatment more than 6 months prior
* At least moderate dyspnea defined by a BDI score of 6 or less in the Self- Administered Computerized Versions of the Baseline and Transition Dyspnea Indexes(SAC-BDI/TDI)13,14 (This cutoff score is close to the score of 5.7 used to define "moderate dyspnea" in the publication that validated the instrument and is selected by attending physicians in the Pulmonary Service as a good indication of "moderate dyspnea" in clinical practice. A typical person with BDI of 6, for example, would be a 52 year old woman who has to pause when walking because of dyspnea and/or has eliminated doing an activity because of dyspnea).
* Able to safely complete the Six Minute Walk Test (6MWT)15 as per attending physician's clinical judgment.
* Respiratory functions clinically stable for the preceding 3 months and expected to be stable for the next 3 months as determined by project PIs and other Pulmonary Medicine faculty.

Exclusion Criteria:

* Life expectancy less than 6 months
* Any cause of dyspnea that is determined by the investigators as readily reversible by other means (e.g. pleural effusion, pulmonary embolism, acute infection, anemia Hb<9.0, etc.)
* Non-English speaking

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
the feasibility | 2 years
  of a breath training program Feasibility is defined by the combination of acceptance rate (number of patients agreeing to participate divided by total number of offered participation), completion rate (percentage of patients completing 75% of practice sessions and providing data on the SAC-BDI/TDI at baseline and 6 weeks) and estimated effect size (20% improvement in SAC-BDI).

CONTACTS AND LOCATIONS:
Overall Officials: Gary Deng, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/